CLINICAL TRIAL: NCT05043727
Title: Effects of Exer Gaming on Balance and Gait in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/2024 Shahbaz
Record Dates: First submitted 2021-08-27; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease; Balance
Keywords: Postural instability,; Parkinson Disease,; Exer Game
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: each participant will be requested to draw either number one or two from box. Group number one will receive exer gaming treatment plan Each Patient received twenty four sessions. Each treatment session will of 50 minutes with two minutes rest between each exercise. Group two will receive conventional treatment plan which will include balance training, gait training, stretching and strengthening exercises.Treatment session will be of 50 minutes with 2 minutes rest period between each exercise.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exer gaming treatment plan (Experimental): Exer gaming treatment plan
  Interventions: Combination Product: Exer gaming
- conventional treatment plan (Active Comparator): conventional treatment plan
  Interventions: Combination Product: conventional treatment plan

INTERVENTIONS:
Combination Product: Exer gaming — exer gaming treatment plan will include perfect ten balance, wii skiing, wiicycling. Each Patient will receive twenty four sessions. Each treatment session was of 50 minutes with two minutes rest between each exercise.
  Arms: Exer gaming treatment plan
Combination Product: conventional treatment plan — it will receive conventional treatment plan which includes balance training, gait training, stretching and strengthening exercises.Each patient will receive twenty four sessions of conventional physical therapy. Treatment session will be of 50 minutes with 2 minutes rest period between each exercise.
  Arms: conventional treatment plan

SUMMARY:
To compare the effects of exer-gaming with conventional physiotherapy on balance and gait in Parkinson's patients

DETAILED DESCRIPTION:
Parkinsons Disease is a progressive neuro degenerative disorder manifested by a broad spectrum of motor and non-motor features. Approximately 500 000 people suffer from Parkinson's Disease in the United States and there are approximately 50,000 new cases reported annually . Postural instability, impaired gait, and freezing episodes are all common occurrences in Parkinson's. Agility activities, including supine-to-stand, ambulation, turning, and reaching activities, have been used to reduce freezing episodes, particularly in the early stages of disease.

Conventional physical therapy(balance training, stretching and strengthening exercises) being used for the balance and gait training in Parkinson. In recent time, there has been development in such treatment plan. Virtual reality based games have been used for such purposes. This study will look at the effects of virtual reality gaming in patients suffering from Parkinson's disease and its outcomes in term of gait and balance training. A randomized clinical trial will be performed. total 16 patients will be included in the study and will be divided into two groups. VR Group will be receiving virtual reality based exercise plan while the CONVENTIONAL group will receive conventional physical therapy . Division will be done through lottery method. Unified parkinson's disease rating scale and dynamic gait index will be used to collect the data. Treatment frequency will be three days per week for three months .

ELIGIBILITY:
Inclusion criteria:

* Diagnosed Parkinson's disease patients in stage I, II,III according to Hoeh n-Yahr classification.
* Patients with balance and gait disorders

Exclusion criteria:

* Other neurological conditions (stroke, Alzheimer)
* Red flag signs (tumors, fractures, infections etc)
* Uncontrolled hypertension.
* Patients with visual disturbances
* Patients with cognitive disorders

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-06 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's diseaserating scale (UPDRS) | 50 minutes
  this test is specifically used in Parkinson patients to check balance

SECONDARY OUTCOMES:
dynamic gait index. | 50 minutes
  to check dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: zeest hashmi, MS NMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao YY, Yang YR, Cheng SJ, Wu YR, Fuh JL, Wang RY. Virtual Reality-Based Training to Improve Obstacle-Crossing Performance and Dynamic Balance in Patients With Parkinson's Disease. Neurorehabil Neural Repair. 2015 Aug;29(7):658-67. doi: 10.1177/1545968314562111. Epub 2014 Dec 24. PMID 25539782
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Lee RG, Tonolli I, Viallet F, Aurenty R, Massion J. Preparatory postural adjustments in parkinsonian patients with postural instability. Can J Neurol Sci. 1995 May;22(2):126-35. doi: 10.1017/s0317167100040208. PMID 7627914